CLINICAL TRIAL: NCT06253793
Title: Tool for Evaluating the Effectiveness of the DENVER Protocol for Attention to Faces (Face) and the Development of Social Communication (Com) in Young Children With Autism Spectrum Disorder (ASD)
Brief Title: Tool for Evaluating the Effectiveness of the DENVER Protocol
Acronym: FACECOM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0401
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Communication; Language; Attention; Face; Children
MeSH Terms: conditions — Autism Spectrum Disorder; Communication; Language; Facies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ASD Experimental group: Children with Autism Spectrum Disorder (ASD) enrolled in the DENVER protocol. Same chronological age (1.5 years to 5 years of age) than children with ASD NOT enrolled in the DENVER protocol. Those children will be recruited and tested at the Alps-Isere Hospital Center (Saint-Egreve, France)
- ASD Control group: Children with Autism Spectrum Disorder (ASD) en NOT enrolled in the DENVER protocol. Same chronological age (1.5 years to 5 years of age) than children with ASD enrolled in the DENVER protocol. Those children will be recruited and tested at the Savoie Hospital Center (Chambery, France) and at the Grenoble University Hospital (Grenoble, France).
- TD control group: Typically developing (TD) children with the same developmental age than children with ASD. Those children will be recruited and tested at the University Grenoble Alps (Grenoble, France).

SUMMARY:
Early remediation of the communicative and social difficulties of children with autism spectrum disorders (ASD) is central. However, from the age of 6-8 months, children with ASD show a lack of attention to social stimuli such as faces: such early avoidance behavior could be at the root of later communicative difficulties (language, attention). The Denver program aims to stimulate social communication and attention to faces in children with ASD aged between 18 and 60 months. Although the Denver protocol is currently recommended by the French National Authority for Health (HAS), the Denver protocol has not yet been widely used or evaluated in France, mainly due to a lack of tools adapted to non-verbal populations. The goal of FaceCom is to help clinicians to evaluate the efficiency of the Denver Protocol.

DETAILED DESCRIPTION:
Early remediation of the communicative and social difficulties of children with autism spectrum disorders (ASD) is central. However, from the age of 6-8 months, children with ASD show a lack of attention to social stimuli such as faces: such early avoidance behavior could be at the root of later communicative difficulties (language, attention). The Denver program aims to stimulate social communication and attention to faces in children with ASD aged between 18 and 60 months. Although the Denver protocol is currently recommended by the French National Authority for Health (HAS), the Denver protocol has not yet been widely used or evaluated in France, mainly due to a lack of tools adapted to non-verbal populations. The goal of FaceCom is to help clinicians to evaluate the efficiency of the Denver Protocol.

For children with ASD benefiting from the Denver protocol, the investigators hypothesize that an improvement in attention to social stimuli (faces, language) should be observed thanks to the Denver protocol intervention. Before the protocol, language and attention to faces of children with ASD included in the Denver protocol should resemble that of children with ASD of the same age who had not benefited from the Denver program. At the end of the Denver protocol, performance from children with ASD included in the Denver protocol should tend towards that of typically developing children of the same developmental age.

ELIGIBILITY:
Inclusion criteria for all groups

* native language: French
* oral consent of the child, if able to do so, written consent of 2 parents or legal guardians

Inclusion criteria for the ASD experimental and control groups:

-ASD Diagnosis The diagnosis of ASD is clinical and is made by the referring physician. It is based on the DSM 5 and the clinical assessment of each patient.

Inclusion criteria for the ASD experimental group:

* absence of neurological pathology (epilepsy, etc.) and known genetic syndrome on admission
* written consent of 2 parents or legal guardians

Non-inclusion criteria for all children:

- primary hearing and visual impairment (unless fully corrected).

Non-inclusion criteria for DT children only:

- a known neurodevelopmental, neurological or psychiatric disorder.

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ASD Experimental Group Children with Autism Spectrum Disorder (ASD) enrolled in the DENVER protocol. Same chronological age (1.5 years to 5 years of age) than children with ASD NOT enrolled in the DENVER protocol.
  ASD Control Group Children with Autism Spectrum Disorder (ASD) NOT enrolled in the DENVER protocol.
  TD Control Group Typically developing (TD) children with the same developmental age than children with ASD
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-05-13 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
looking time during natural social scenes | measure of 10 minutes :once for the ASD control and TD control groups. Repeated 4 times (every 3 months) for the ASD Experimental group
  Looking time in natural interaction situations is measured by recording the direction and time of the child's gaze at faces and objects in real social scenes using a video camera. The recording is then viewed by experimenters and manually coded frame by frame (sampling frequency 25 frames/second), determining which areas of interest (face, object) are looked at by the child at each time step. This measurement is less precise than the following one, but enables us to assess these children's social skills in real scenes of adult/child interaction (PART 1 of the data collection).
looking time to social scenes presented on a screen | measure of 10 minutes :once for the ASD control and TD control groups. Repeated 4 times (every 3 months) for the ASD Experimental group
  Looking time during the viewing of social scenes presented on a screen is measured using an eye-tracking system, suitable for studying populations as young as 3 months. The eye-tracker is a device used to measure very precisely (x and y spatial coordinates at a temporal sampling frequency of around 30 Hertz) where the child's gaze rests and for how long in a 2D social scene presented on screen (PART 2 of data collection). These data are collected automatically by the eye tracker (spatial coordinates at each time step) and then coded into areas of interest (gaze locations: eyes, mouth...).

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde FORT, PhD, Study Chair — University Grenoble Alps; Isabelle Palacios, MD, Study Chair — Alps-Isere Hospital Center
Locations (3):
- France (3):
  - Alps-Isere Hospital Center, Saint-Égrève, Isere
  - Savoie Hospital Center, Chambéry, Savoie
  - University Grenoble Alps, Grenoble

IPD SHARING:
Plan to Share IPD: No